CLINICAL TRIAL: NCT07253779
Title: The Effect of Mentoring Programme on Reality Shock, Clinical Adaptation and Professional Competencies of New Graduated Nurses
Brief Title: The Effect of a Mentoring Program for New Graduate Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Selma Karakaplan, Registered Nurse (RN), Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IUCFNHF
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Nurse Education
Keywords: Mentoring Programme; Reality Shock; Clinical Adaptation; Professional Competence

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group, which received the mentoring program, or the control group, which did not receive any intervention. Randomization was conducted using unique participant codes and random numbers generated via www.random.org to ensure allocation concealment. Data were collected at three time points: before the intervention, immediately after the intervention, and three months later. This pretest-posttest control group design allowed for comparison of changes over time between the two groups.
  This study did not involve any patients, drugs, or medical devices. It focused solely on a professional mentoring intervention for newly graduated nurses.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentoring programme group (Experimental): The intervention group participated in a structured, four-week behavioral mentoring program. Mentors and mentees worked together in regular training and support sessions. Participants were assessed at three time points: before the program, immediately after the program, and three months post-intervention to evaluate changes in clinical adaptation, reality shock, and professional competence.
  Interventions: Behavioral: Mentoring Programme
- No Intervention (No Intervention): The control group did not receive the mentoring program. Participants continued with the standard orientation and support provided by the hospital. They were assessed at the same three time points as the intervention group to allow comparison of clinical adaptation, reality shock, and professional competence.

INTERVENTIONS:
Behavioral: Mentoring Programme — A structured, four-week behavioral mentoring program developed for newly graduated nurses. During the program, mentors and mentees worked together through regular training and support sessions designed to enhance clinical adaptation, reduce reality shock, and improve professional competence. Mentors provided individualized guidance, feedback, and educational support throughout the process. Participants were assessed before the intervention, immediately after, and three months post-intervention to evaluate changes in the outcomes.
  Arms: Mentoring programme group

SUMMARY:
The study was conducted to evaluate the effects of mentoring programme on the reality shock, clinical adaptation, and professional competence of new graduate nurses. The research questions were: Are the reality shock scores of new graduate nurses participating in the mentoring program lower than those in the control group? Is the clinical adaptation of new graduate nurses participating in the mentoring program higher than those in the control group? Are the professional competence scores of new graduate nurses participating in the mentoring program higher than those in the control group? The study was a mixed-use study with intervention and control groups, blinded design, randomized controlled experimental method, and focus group interview method. The number of nurses comprising the sample was determined using power analysis. The study population consisted of 65 newly graduated nurses who had started the institution, and the sample consisted of 56 nurses (28 in the intervention group and 28 in the control group) who were randomly assigned. In the first phase of the study, mentor nurses were trained according to the developed training program, and in the second phase, the mentor nursing practice was implemented. During this period, nurses in the control group received a one-month routine clinical orientation training, nurses in the intervention group received a one-month nursing mentorship program, and newly graduated nurses were monitored for three months. Quantitative data were collected before and after the nursing mentorship program, and in the third month of the study. Focus Group Interviews were conducted before and after the nursing mentorship program to collect qualitative data.

DETAILED DESCRIPTION:
This study evaluated the effect of a mentoring program on reality shock, clinical adaptation, and professional competence of new graduate nurses. Participants were randomly assigned to either the intervention group, which received the mentoring program, or the control group, which did not receive any intervention. Randomization was performed using unique codes and random numbers generated via www.random.org

, ensuring allocation concealment. Outcome measures were collected at three time points: before the intervention, immediately after the intervention, and three months post-intervention.

A qualitative component was conducted using focus group interviews to explore participants' perceptions and experiences regarding the mentoring program. The qualitative data complemented the quantitative measures and provided in-depth insights into the participants' adaptation process. Participants were not informed of their group assignment, and information about the mentoring program was provided in a way that did not break the blinding.

ELIGIBILITY:
Inclusion Criteria:

* New graduate
* First time working as a nurse

Exclusion Criteria:

* Leaving the institution during the research process
* Not having completed the orientation process

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of reality shock in newly graduated nurses | Measured at three time points: baseline (before starting the mentoring program), immediately after the one-month mentoring program, and at three months after program initiation
  Reality shock score :The Reality Shock scale was used for this measurement. It is an assessment tool developed by Cennet Çiriş Yıldız and Yasemin Ergün in 2019 to determine the reality shock of newly graduated nurses. The scale consists of 47 questions and 4 subdimensions. These subdimensions are Collaboration and Relationships (24 items), Professional Knowledge (12 items), Responsibility (7 items), and Performance (4 items). The scale is a 5-point Likert-type scale with scores of Never (1), Rarely (2), Sometimes (3), Often (4), and Always (5). There are no reverse-coded items. The minimum score obtained from the scale is 47, and the maximum is 235. Increasing mean scores on the scale subdimensions indicate an increasing level of reality shock.
Evaluation of professional competencies of newly graduated nurses | Measured at three time points: baseline (before starting the mentoring program), immediately after the one-month mentoring program, and at three months after program initiation
  The Nursing Professional Competency Scale was used for this measurement. This scale is an assessment tool developed by Figen Çalışkan and Emine Şenyuva in 2020 to measure the professional competencies of nurses. The scale consists of 67 items and 7 subdimensions. These subdimensions are Diagnosis, Implementation of the Nursing Process, Health/Patient Education, Professional Development, Ethical Practices, Critical Thinking and Teamwork, and Research and Development. The scale is a 4-point Likert-type scale with scores of Always (4), Usually (3), Sometimes (2), and Never (1). All items on the scale are positive, and there are no reverse-coded items. The minimum score on the scale is 67 and the maximum score is 268. An increase in the scale score indicates an increase in the professional competence of nurses.
Evaluation of clinical adaptation of newly graduated nurses | Measured at three time points: baseline (before starting the mentoring program), immediately after the one-month mentoring program, and at three months after program initiation
  Clinical orientation of new graduate nurses was assessed using the Clinical Orientation Portfolio. This measurement tool was developed by the researcher to assess the clinical orientation of new graduate nurses and the competencies they should possess. The Clinical Orientation Portfolio consists of seven competency areas and 30 competency statements.
Evaluation of new graduate nurses' experiences and perceptions regarding the mentoring program | Assessed before the mentoring program and immediately after its completion
  A focus group interview form was used for this measurement. To assess new graduate nurses' views on the mentoring program, the first interview consisted of four items, and the final interview consisted of a semi-structured questionnaire consisting of five main items and sub-items. Care was taken to ensure that the questions were structured to allow for sub-questions to be asked during the interview if necessary, were clear and simple enough to be easily understood, and were not directive. Before the data collection phase, a preliminary interview was conducted with a group of eight individuals excluded from the sample, and the focus group interview questions were tested and finalized.

CONTACTS AND LOCATIONS:
Overall Officials: Selma Karakaplan, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Dr. Lütfi Kırdar City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality and ethical considerations. Only aggregated results will be reported.

REFERENCES:
- See also: Nursing professional competence scale — https://bakirkoymedj.org/articles/doi/BMJ.galenos.2021.2021.11-2